CLINICAL TRIAL: NCT05626855
Title: An Open-Label, Multicenter, Extension Trial to Evaluate the Long-Term Safety and Efficacy of Apitegromab in Patients With Type 2 and Type 3 Spinal Muscular Atrophy Who Completed Previous Investigational Trials of Apitegromab
Brief Title: Long-Term Safety & Efficacy of Apitegromab in Patients With SMA Who Completed Previous Trials of Apitegromab
Acronym: ONYX
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Scholar Rock, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRK-015-004
Record Dates: First submitted 2022-11-07; First posted 2022-11-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Spinal Muscular Atrophy; Spinal Muscular Atrophy Type 3; Spinal Muscular Atrophy Type 2; SMA; Neuromuscular Diseases; Muscular Atrophy; Atrophy; Muscular Atrophy, Spinal; Neuromuscular Manifestations; Anti-myostatin
MeSH Terms: conditions — Muscular Atrophy, Spinal; Spinal Muscular Atrophies of Childhood; Neuromuscular Diseases; Muscular Atrophy; Atrophy; Neuromuscular Manifestations | interventions — apitegromab

STUDY DESIGN:
Intervention Model Description: Open Label Extension Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Period (Experimental): Patients who are ≥2 years of age with Type 2 and Type 3 SMA will receive apitegromab 20 mg/kg every 4 weeks by intravenous (IV) infusion during the 104-week Treatment Period
  Interventions: Drug: Apitegromab

INTERVENTIONS:
Drug: Apitegromab — Apitegromab (SRK-015) is an investigational, fully human immunoglobulin G4 monoclonal antibody that specifically binds to human proforms (i.e., inactive precursor forms) of myostatin, pro- and latent- myostatin, with high affinity, inhibiting activation of myostatin, a negative regulator of muscle growth and strength.

SUMMARY:
The ONYX study is an Open-Label, Multicenter, Extension study that will evaluate the long-term safety and efficacy of Apitegromab in Patients with Type 2 and Type 3 SMA who have completed TOPAZ or SAPPHIRE.

ELIGIBILITY:
Inclusion Criteria:

* Patients have completed the Phase 2 TOPAZ (Study SRK-015-002) trial or the Phase 3 SAPPHIRE (Study SRK-015-003) trial. (For TOPAZ, completed is defined as completion of Visit EC14 in Extension Period C or participating in TOPAZ at the time the trial is ended. For SAPPHIRE, completed is defined as completion of Visit 14 or participating in SAPPHIRE at the time the trial is ended)
* Estimated life expectancy >2 years from the Baseline Visit (Day 1)
* Able to receive study drug infusions and provide blood samples through the use of a peripheral IV or a long-term IV access device that the patient has placed for reasons independent from the trial
* Able to adhere to the requirements of the protocol, including travel to the trial site and completing all trial procedures and trial visits
* Females of childbearing potential must have a negative pregnancy test at the Baseline Visit and agree to use at least 1 highly effective method of contraception throughout the trial and for 20 weeks after the last dose of apitegromab

Exclusion Criteria:

* Patient permanently discontinued study treatment during the feeder trial (i.e., TOPAZ or SAPPHIRE)
* Nutritional status that was not stable over the past 6 months and is not anticipated to be stable throughout the trial or medical necessity for a gastric/nasogastric feeding tube, where the majority of feeds are given by this route, as assessed by the Investigator
* Patient is currently enrolled in any investigational drug trial other than TOPAZ or SAPPHIRE
* Prior history of severe hypersensitivity reaction or intolerance to SMN-targeted therapies
* Prior history of severe hypersensitivity reaction or intolerance to apitegromab
* Use of chronic daytime noninvasive ventilatory support for >16 hours daily in the 2 weeks before dosing, or anticipated to regularly receive such daytime ventilator support chronically throughout the trial
* Any acute or comorbid condition interfering with the well-being of the patient at the patient's last visit in TOPAZ or SAPPHIRE, (including active systemic infection, the need for acute treatment, or inpatient observation due to any reason). After resolution of the condition, the patient can be enrolled in the trial if they meet all the other eligibility criteria.
* Pregnant or breastfeeding
* Any other condition or clinically significant laboratory result or ECG value that, in the opinion of the Investigator, may compromise safety or compliance, would preclude the patient from successful completion of the trial, or interfere with the interpretation of the results

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2029-05-02 (Estimated)

PRIMARY OUTCOMES:
Evaluate the long-term safety and tolerability of apitegromab in patients with Type 2 and Type 3 SMA | Up to 6 years
  Incidence of TEAEs and SAEs by severity

SECONDARY OUTCOMES:
Evaluate the long-term efficacy of apitegromab by assessing changes in motor function outcome measures at prespecified time points | Up to 6 years
  Hammersmith Functional Motor Scale Expanded (HFMSE) total score at prespecified time points (excludes ambulatory patients)
Evaluate the long-term efficacy of apitegromab by assessing changes in motor function outcome measures at prespecified time points | Up to 6 years
  Revised Upper Limb Module (RULM) total score at prespecified time points (excludes ambulatory patients)
Evaluate the long-term efficacy of apitegromab by assessing changes in motor function outcome measures at prespecified time points | Up to 6 years
  Number of World Health Organization (WHO) motor development milestones attained at prespecified time points (excludes ambulatory patients)
Evaluate the long-term efficacy of apitegromab by assessing changes in motor function outcome measures at prespecified time points | Up to 6 years
  Revised Hammersmith Scale (RHS) total score
Evaluate the long-term efficacy of apitegromab by assessing changes in motor function outcome measures at prespecified time points | Up to 6 years
  Results for 6-Minute Walk Test
Evaluate the long-term efficacy of apitegromab by assessing changes in motor function outcome measures at prespecified time points | Up to 6 years
  30-Second Sit-to-Stand
Further evaluate the immunogenicity of apitegromab | Up to 6 years
  Presence or absence of antidrug antibody (ADA) against apitegromab in serum from blood samples

OTHER OUTCOMES:
Further characterize the PK of apitegromab | Up to 6 years
  Apitegromab concentrations in serum from blood samples at prespecified time points
Further evaluate the pharmacodynamic (PD) effects of apitegromab | Up to 6 years
  Total latent myostatin concentrations in blood samples at prespecified time points
To further evaluate the effect of apitegromab on patient/caregiver-reported disability, and fatigability. | Up to 6 years
  Pediatric Evaluation of Disability Inventory Computer Adaptive Test (PEDI-CAT) at prespecified time points
To further evaluate the effect of apitegromab on patient/caregiver-reported disability, and fatigability. | Up to 6 years
  Patient-reported Outcomes Measurement Information System (PROMIS) Fatigue Questionnaire at prespecified time points
To further evaluate the effect of apitegromab on patient/caregiver-reported disability, and fatigability. | Up to 6 years
  Assessment of Caregiver Experience with Neuromuscular Disease (ACEND) at prespecified time points

CONTACTS AND LOCATIONS:
Locations (49):
- United States (25):
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - UCSD Altman Clinical and Translational Research, La Jolla, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Stanford Neuroscience Health Center, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Nemours Biomedical Research, Orlando, Florida
  - Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Fairway, Kansas
  - Johns HopkinsHospital, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Gillette Children's Specialty Healthcare, Saint Paul, Minnesota
  - Washington University Medical Campus, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - University of Texas Southwestern - Pediatric Neurology, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - Children's Specialty Group PLLC (Children's Hospital of The King's Daughters), Newport News, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - University of Wisconsin Hospital, Madison, Wisconsin
- Belgium (3):
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
  - CHR Citadelle, Liège
- France (3):
  - CHRU de Lille - Hpital Jeanne de Flandre, Lille
  - Hopital Trousseau - I-Motion, Paris
  - CHU Toulouse Hopital des Enfants, Toulouse
- Germany (4):
  - Universitätskinderklinik Bonn, Abteilung für Neuropädiatrie und SPZ, Bonn
  - Universitatsklinikum Essen, Essen
  - Universitatsklinikum Freiburg, Freiburg im Breisgau
  - Klinikum der Universitat Munchen, Dr. von Haunersches Kinderspital, Abteilung fur Kinderneurologie und Entwicklungsneurologie, Munchen, Bayern
- Italy (5):
  - Istituto Giannina Gaslini, Centro Traslazionale di Miologia e Patologie Neurodegenerative, Genova
  - UOC NEUROLOGIA E MALATTIE NEUROMUSCOLARI A.O.U Policlinico G. Martino, Messina
  - Carlo Besta Neurological Research Institute, Milan
  - NeuroMuscular Omnicentre, Milan
  - Fondazione Policlinico Universitario A. Gemelli, Roma
- UMC Utrecht, Utrecht, Netherlands
- Poland (3):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Oddział Kliniczny Neurologii Dzieci i Młodzieży, Poznan
  - Instytut Pomnik - Centrum Zdrowia Dziecka, Warsaw
- Spain (2):
  - Hospital Sant Joan de Deau, Barcelona
  - Hospital Universitari i Politecnic La Fe, Valencia
- United Kingdom (3):
  - Leeds Children's Hospital Clinical Research, Leeds
  - Great Ormond Street Hospital for Children, London
  - University of Oxford, Oxford

IPD SHARING:
Plan to Share IPD: No